CLINICAL TRIAL: NCT04494529
Title: Single Dose Antenatal Corticosteroids (SNACS) Pilot Randomized Control Trial for Women at Risk of Preterm Birth
Brief Title: Single Dose Antenatal Corticosteroids (SNACS) for Women at Risk of Preterm Birth
Acronym: SNACS Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sarah McDonald, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SNACS Pilot Trial
Record Dates: First submitted 2020-07-16; First posted 2020-07-31 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Preterm Birth; Complication of Prematurity; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications
Keywords: Premature birth; Preterm birth; Obstetric labor; Betamethasone Valerate; Betamethasone-17,21-dipropionate; Betamethasone benzoate; Betamethasone sodium phosphate; Anti-Inflammatory Agents; Glucocorticoids; Hormones; Hormone Substitutes; Hormone Antagonists; Physiological Effect of Drugs; Anti-Asthmatic Agents; Respiratory System Agents
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications | interventions — Betamethasone

STUDY DESIGN:
Intervention Model Description: Pilot double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-Dose (12 mg betamethasone + placebo) (Placebo Comparator): The standard course of betamethasone consists of 2 intramuscular injections of 12 mg betamethasone 24 hours apart for a total dose of 24 mg. Before enrolment and randomization in the SNACS trial, all women will have received a first 12 mg injection of betamethasone according to local hospital protocols. After this first injection, randomization is performed.
  Participants randomized to the experimental "Single-Dose" arm will receive a similar appearing placebo injection instead of the standard 2nd dose of 12 mg of betamethasone (i.e. they will receive the experimental single-dose regimen, total 12 mg of betamethasone only from the first injection).
  Interventions: Drug: 12 mg betamethasone + placebo
- Double-Dose (12 mg betamethasone + 12 mg betamethasone) (Active Comparator): The standard course of betamethasone consists of 2 intramuscular injections of 12 mg betamethasone 24 hours apart for a total dose of 24 mg. Before enrolment and randomization in the SNACS trial, all women will have received a first 12 mg injection of betamethasone according to local hospital protocols. After this first injection, randomization is performed.
  Participants randomized to the "Double-Dose" arm will receive the standard 2nd dose of 12 mg of betamethasone injected intramuscularly (i.e. they will receive the standard double-dose regimen, total 24 mg of betamethasone).
  Interventions: Drug: 24 mg betamethasone

INTERVENTIONS:
Drug: 12 mg betamethasone + placebo — After the first intramuscular injection of 12 mg of betamethasone, participants randomized to the "Placebo Comparator" group will receive 1 intramuscular injection of placebo.
  Arms: Single-Dose (12 mg betamethasone + placebo)
Drug: 24 mg betamethasone — After the first intramuscular injection of 12 mg of betamethasone, participants randomized to the "Active Comparator" group will receive the standard 2nd intramuscular injection of 12 mg of betamethasone.
  Arms: Double-Dose (12 mg betamethasone + 12 mg betamethasone)

SUMMARY:
Antenatal corticosteroids (ACS) reduce the risks of neonatal death and morbidities, such as respiratory distress syndrome, in preterm infants.

Standard of care for women at risk of preterm birth includes 2 doses of 12 mg betamethasone (for a total of 24 mg) to accelerate fetal lung maturity.

We plan to conduct a pilot clinical trial to determine the feasibility of a trial comparing half the usual dose (total 12 mg) of betamethasone to the standard double dose (total 24 mg) of betamethasone.

The results of this pilot will be combined with the full-scale RCT (NCT05114096) for which we have received funding from the Canadian Institutes of Health Research (CIHR).

DETAILED DESCRIPTION:
Preterm infants are at risk of mortality and morbidity. Antenatal corticosteroids (ACS) reduce the risks of neonatal death and morbidities, such as respiratory distress syndrome.

Standard of care for women at risk of preterm birth includes 2 doses of 12 mg betamethasone (for a total of 24 mg) to accelerate fetal lung maturity. There are no published clinical trial data on the benefits or risks of a single dose of antenatal corticosteroid vs. standard double doses.

Pilot trials are now viewed as an "almost essential prerequisite" to large, expensive, full scale studies. Thus, we plan to conduct a pilot clinical trial to determine the feasibility of a trial comparing half the usual dose (12 mg of betamethasone + placebo) to the standard double dose (12 mg + 12 mg of betamethasone), as well as the feasibility of the study protocol. Secondary outcomes will include process outcomes and pilot clinical outcomes, that will be combined with the full-scale RCT for which we have received funding from CIHR.

We plan to conduct a 24-month corrected gestational age follow-up, which will consist principally of 2 validated parent-filled questionnaires:

1. Ages and Stages Questionnaire-3 (ASQ)
2. Child Behavior Checklist
3. A single question parent report of whether there has been a physician diagnosis of cerebral palsy. (recommended by our parent partners)

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women at risk of preterm birth with a singleton or twins between =>22+0/7 and <=34+6/7 weeks' gestation
2. Pregnant with either singletons or twins
3. Has already received the first dose of 12 mg intramuscular betamethasone within the past 24 hours
4. All fetuses are alive and without compromise as per ultrasound or fetal heart monitor
5. Is capable of giving informed, written consent in English

Exclusion Criteria:

1. Any contraindications to receiving corticosteroids
2. Requires chronic doses of corticosteroids secondary to a medical condition (e.g. systemic lupus erythematosus, severe asthma, congenital adrenal hyperplasia, etc.)
3. Received any prior doses of antenatal corticosteroids except for the 1st dose of 12 mg intramuscular betamethasone
4. Had any previous participation in this trial
5. Pregnant with a fetus with severe congenital anomaly (e.g. anencephaly, transposition of the great arteries, etc.) or major chromosomal abnormalities (e.g. Trisomy 18, Trisomy 21, etc.)
6. Pregnant with monoamniotic/monochorionic (Mono/Mono) twins

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a full-scale trial | 5-6 months
  Feasibility of conducting a full-scale trial will be defined as => 50% recruitment of approached participants
Feasibility of the study protocol | 5-6 months
  Feasibility of the study intervention will be defined as => 98% compliance with the protocol

SECONDARY OUTCOMES:
Process outcomes | 5-6 months
  The proportions of patients who: will be approached by the circle of care, and will agree to be approached by the research team, and will agree to participate
Neonatal mortality rates | 5-6 months
  Pilot clinical data on neonatal mortality, from medical records
Respiratory morbidity rates | 5-6 months
  Pilot clinical data on respiratory morbidity, from medical records
Severe intraventricular haemorrhage rates | 5-6 months
  Pilot clinical data on severe intraventricular haemorrhage, from medical records
Rates of severe bowel problems due to necrotizing enterocolitis | 5-6 months
  Pilot clinical data on severe bowel problems due to necrotizing enterocolitis, from medical records
Duration of mechanical ventilation requiring an endotracheal tube | 5-6 months
  Pilot clinical data on duration of mechanical ventilation requiring an endotracheal tube, from medical records
Need for supplemental oxygen and duration | 5-6 months
  Pilot clinical data on need for supplemental oxygen and duration, from medical records
Late respiratory morbidity (i.e. bronchopulmonary dysplasia) rates | 5-6 months
  Pilot clinical data on late respiratory morbidity (i.e. bronchopulmonary dysplasia), from medical records
Early neonatal sepsis rates | 5-6 months
  Pilot clinical data on early neonatal sepsis, from medical records
Severe late brain injury (periventricular leukomalacia) rates | 5-6 months
  Pilot clinical data on severe late brain injury (periventricular leukomalacia), from medical records
Intrauterine fetal demise rates | 5-6 months
  Pilot clinical data on intrauterine fetal demise, from medical records
Duration of ventilatory support not requiring an endotracheal tube | 5-6 months
  Pilot clinical data on duration of ventilatory support not requiring an endotracheal tube, from medical records
Rates of hypotension < 48 hours of life requiring treatment with hydrocortisone or inotropic medications | 5-6 months
  Pilot clinical data on hypotension < 48 hours of life requiring treatment with hydrocortisone or inotropic medications, from medical records
Length of stay in neonatal intensive care unit | 5-6 months
  Pilot clinical data on length of stay in neonatal intensive care unit, from medical records
Anthropometry composite (<10% of expected weight, length, or head circumference for birth week) | 5-6 months
  Pilot clinical data on anthropometry (<10% of expected weight, length, or head circumference for birth week), from medical records
Number of infants with retinopathy of prematurity needing treatment | 5-6 months
  Pilot clinical data on retinopathy of prematurity needing treatment, from medical records
Patent ductus arteriosus needing a closure procedure | 5-6 months
  Pilot clinical data on number of infants with patent ductus arteriosus needing a closure procedure, from medical records
24-month follow-up | 18-30 months
  Neurosensory/developmental progress at 24 months corrected gestational age, which will consist principally of 2 validated parent-filled questionnaires:
  1. Ages and Stages Questionnaire-3 (ASQ)
  2. Child Behavior Checklist
  3. A single-question parent report of whether there has been a physician diagnosis of cerebral palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D McDonald, MD, MSc, FRCSC, Principal Investigator — McMaster University; Kellie Murphy, MD, MSc, FRCSC, Principal Investigator — University of Toronto
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No